CLINICAL TRIAL: NCT01216111
Title: A Prospective， Randomized， Open-label， Multicentric，phaseIII Clinical Trial Compared With PC and CEF100 Followed by Docetaxel as Adjuvant Chemotherapy Regimen for Chinese Primary Triple Negative Breast Cancer Patients
Brief Title: Adjuvant Platinum and Taxane in Triple-negative Breast Cancer (PATTERN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Chinese Anti-Cancer Association (Other)
Responsible Party: Principal Investigator, Zhimin Shao, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan TNBC Adjuvant CT
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Triple Negative Breast Cancer
Keywords: triple negative breast cancer，local recurrence,distant metastasis
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — TP protocol; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6 cycles of PC adjuvant chemotherapy (Experimental): paclitaxel 80 mg/m2 and carboplatin (area under the curve [AUC]= 2) on day 1, 8, 15 every 28 days for six cycles
  Interventions: Drug: Paclitaxel Cisplatin
- 3 cycles of FEC followed by 3 cycles of Docetaxel (Active Comparator): fluorouracil 500 mg/m2, epirubicin 100 mg/m2, and cyclophosphamide 500 mg/m2 intravenously on day 1 every 21 days for three cycles followed by docetaxel 100 mg/m2 intravenously
  Interventions: Drug: fluorouracil epirubicin cyclophosphamide and docetaxel (FEC-T)

INTERVENTIONS:
Drug: Paclitaxel Cisplatin — Paclitaxel 80 mg/m2 D1，8，15 Cisplatin AUC=2 D1，8，15
  1 cycle = 28days
  PC*6
  Arms: 6 cycles of PC adjuvant chemotherapy
Drug: fluorouracil epirubicin cyclophosphamide and docetaxel (FEC-T) — fluorouracil 500 mg/m2, epirubicin 100 mg/m2, and cyclophosphamide 500 mg/m2 intravenously on day 1 every 21 days for three cycles followed by docetaxel 100 mg/m2 intravenously
  Arms: 3 cycles of FEC followed by 3 cycles of Docetaxel

SUMMARY:
Previous studies in Western country show that triple-negative breast cancer has aggressive clinical and pathological features compared with non-triple negative breast cancer, including onset at a young age, advanced clinical stage, high histologic and nuclear grade and more distant recurrence.

According to the characteristics of triple negative breast tumor, the TNBC patients can benefit neither from hormonal therapies nor from target therapies against Her2 receptors. The only systemic therapy currently available is chemotherapy, and prognosis remains poor. It becomes more and more important to investigate the sensitive chemotherapy regimen for triple negative patients.

Cisplatin-based regimen was active for the patients of lung cancer, colorectal cancer and ect. Triple negative breast cancer patients were more sensitive to platinum-based chemotherapy regimens according to the results of some retrospective studies.

The investigators hypothesized that paclitaxel combined with cisplatin is more sensitive to triple negative breast cancer compared with CEF followed by docetaxel.

DETAILED DESCRIPTION:
Eligibility Female adults(18-70 years old) are eligible if they had histologically confirmed primary breast cancer. Patients also had Eastern Cooperative Oncology Group(ECOG) Performance status of 0 or 1, absolute neutrophil count (ANC)>1500/mm3,hemoglobin >90g/dL, and platelet count >100,000/mm3,creatinine<2.5 times the upper limit of normal(ULN)）, transaminases<3 times ULN or alkaline phosphatase<4 times ULN if transaminases was normal, and total bilirubin <1.5 times ULN. Exclusion criteria were active infection, pregnancy, other primary malignancy (except in situ carcinoma of cervix or adequately treated nonmelanomatous carcinoma of the skin), any documented distant metastasis and uncontrolled systemic diseases.

This study protocol was approved by institutional ethic review boards and conducted according to guidelines for good clinical practice and the Helsinki Declaration.All patients provided written informed consent.

Outcome Measures Primary Endpoint：5 year Disease Free Survival（DFS） Second Endpoints：5 year distant disease free survival （DDFS） 5 year event free survival （EFS） 5 year overall survival （OS） 5 year DFS in gBRCA1 mutation carriers and homologous recombination repair (HRR)-related gene mutation carriers

ELIGIBILITY:
Inclusion Criteria:

1. Women aged from 18 to 70 years;
2. Histologically proven invasive unilateral breast cancer (regardless of the type);
3. Initial clinical condition compatible with complete initial resection;
4. No residual macro or microscopic tumor after surgical excision;
5. Beginning of chemotherapeutic treatment no later than day 42 after the initial surgery;
6. positive lymph node or negative lymph node with tumor size > 1.0cm
7. Patient presenting one of the following criteria (reviewed before randomization by referent pathologist):

   Triple negative （ER-PR-Her-2-） Hormone receptor negativity is defined as ER<1%, PR<1% (IHC), HER2 negativity is defined as IHC 0-1+, or [IHC 2+ and FISH or CISH negative].
8. No clinically or radiologically detectable metastases (M0);
9. No peripheral neuropathy > 1;
10. WHO Performance status (ECOG) of 0 or 1;
11. Adequate recovery from recent surgery (at least one week must have elapsed from the time of a minor surgery (excluding breast biopsy); at least three weeks for major surgery);
12. Adequate hematological function (neutrophil count ³ 2x109/l, platelet count ³ 100x 109/l, Hemoglobin > 9 g/dl);
13. Adequate hepatic function: ASAT and ALAT ≤ 3 ULN alkaline phosphatases ≤ 2.5 ULN,total bilirubin ≤ 1,5 ULN;
14. Adequate renal function: serum creatinine ≤ 1 ULN;
15. Patients accepting contraception intake during the overall length of treatment if of childbearing potential;
16. Adequate cardiac function, LEVF value > 50% by Muga scan or echocardiography;
17. Signed written informed consent.

Exclusion Criteria:

1. Bilateral breast cancer or patient with controlateral DCIS;
2. Any metastatic impairment, including homolateral sub-clavicular node involvement,regardless of its type;
3. Any T4 lesion (UICC1987) (cutaneous invasion, deep adherence, inflammatory breast cancer);
4. ER+ or PR+ or Her-2 overexpression
5. Any clinically or radiologically suspect and non-explored damage to the controlateral breast;
6. Any chemotherapy, hormonal therapy or radiotherapy before surgery;
7. Previous cancer (excepted cutaneous baso-cellular epithelioma or uterin peripheral ephitelioma) in the preceding 5 years, including invasive controlateral breast cancer;
8. Patients already included in another therapeutic trial involving an experimental drug;
9. Patients with other concurrent severe and/or uncontrolled medical disease or infection which could compromise participation in the study;
10. LEVF < 50% (MUGA scan or echocardiography);
11. Clinically significant cardiovascular disease (e.g. unstable angina, congestive heart failure, uncontrolled hypertension (>150/90), myocardial infarction or cerebral vascular accidents) within 6 months prior to randomization;
12. Known prior severe hypersensitivity reactions to agents containing Cremophor EL;
13. Women of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and up to 8 weeks after treatment completion;
14. Women who are pregnant or breastfeeding. Adequate birth control measures should be taken during study treatment phase;
15. Women with a positive pregnancy test en enrollment or prior to study drug administration;
16. Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial;
17. Individual deprived of liberty or placed under the authority of a tutor.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 647 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-04-20 (Actual); Study Completion 2016-04-20 (Actual)

PRIMARY OUTCOMES:
disease-free survival | 5 year
  time from random assignment to first relapse (local, regional and distant), contralateral breast cancer

SECONDARY OUTCOMES:
distant disease-free survival | 5 year
  time from random assignment to distant recurrence or death
relapse-free survival | 5 year
  time from the date of randomization to local, regional, distant relapse or death
disease-free survival gBRCA1 mutation carriers and homologous recombination repair (HRR)-related gene mutation carriers | 5 year
overall survival | 5 year
  time from randomization until death with any cause

REFERENCES:
- [Background] Perou CM, Sorlie T, Eisen MB, van de Rijn M, Jeffrey SS, Rees CA, Pollack JR, Ross DT, Johnsen H, Akslen LA, Fluge O, Pergamenschikov A, Williams C, Zhu SX, Lonning PE, Borresen-Dale AL, Brown PO, Botstein D. Molecular portraits of human breast tumours. Nature. 2000 Aug 17;406(6797):747-52. doi: 10.1038/35021093. PMID 10963602
- [Background] Carey LA, Dees EC, Sawyer L, Gatti L, Moore DT, Collichio F, Ollila DW, Sartor CI, Graham ML, Perou CM. The triple negative paradox: primary tumor chemosensitivity of breast cancer subtypes. Clin Cancer Res. 2007 Apr 15;13(8):2329-34. doi: 10.1158/1078-0432.CCR-06-1109. PMID 17438091
- [Background] Yehiely F, Moyano JV, Evans JR, Nielsen TO, Cryns VL. Deconstructing the molecular portrait of basal-like breast cancer. Trends Mol Med. 2006 Nov;12(11):537-44. doi: 10.1016/j.molmed.2006.09.004. Epub 2006 Sep 29. PMID 17011236
- [Background] Reis-Filho JS, Tutt AN. Triple negative tumours: a critical review. Histopathology. 2008 Jan;52(1):108-18. doi: 10.1111/j.1365-2559.2007.02889.x. PMID 18171422
- [Background] Cleator S, Heller W, Coombes RC. Triple-negative breast cancer: therapeutic options. Lancet Oncol. 2007 Mar;8(3):235-44. doi: 10.1016/S1470-2045(07)70074-8. PMID 17329194
- [Background] Dent R, Trudeau M, Pritchard KI, Hanna WM, Kahn HK, Sawka CA, Lickley LA, Rawlinson E, Sun P, Narod SA. Triple-negative breast cancer: clinical features and patterns of recurrence. Clin Cancer Res. 2007 Aug 1;13(15 Pt 1):4429-34. doi: 10.1158/1078-0432.CCR-06-3045. PMID 17671126
- [Background] Hayes DF, Ethier S, Lippman ME. New guidelines for reporting of tumor marker studies in breast cancer research and treatment: REMARK. Breast Cancer Res Treat. 2006 Nov;100(2):237-8. doi: 10.1007/s10549-006-9253-5. Epub 2006 Jun 14. No abstract available. PMID 16773436
- [Derived] Yu KD, Ye FG, He M, Fan L, Ma D, Mo M, Wu J, Liu GY, Di GH, Zeng XH, He PQ, Wu KJ, Hou YF, Wang J, Wang C, Zhuang ZG, Song CG, Lin XY, Toss A, Ricci F, Shen ZZ, Shao ZM. Effect of Adjuvant Paclitaxel and Carboplatin on Survival in Women With Triple-Negative Breast Cancer: A Phase 3 Randomized Clinical Trial. JAMA Oncol. 2020 Sep 1;6(9):1390-1396. doi: 10.1001/jamaoncol.2020.2965. PMID 32789480